CLINICAL TRIAL: NCT01333761
Title: FDS-0004 Cardiox Shunt Detection Technology Study
Brief Title: Cardiox Shunt Detection Technology Study
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: 1)new FDS device design 2)improved Valsalva procedure 3)improved headbands and earpads.
Sponsor: Cardiox Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: FDS-0004
Record Dates: First submitted 2011-03-31; First posted 2011-04-12 (Estimated); Last update posted 2013-01-09 (Estimated); Status verified 2013-01

CONDITIONS: Patent Foramen Ovale
Keywords: right to left cardiac shunt finding
MeSH Terms: conditions — Foramen Ovale, Patent

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TCD/Cardiox FDS/TEE testing (Experimental): All patients enrolled will be evaluated with TCD and Cardiox FDS and TEE for the presence of RTLS.
  Interventions: Device: Cardiox FDS

INTERVENTIONS:
Device: Cardiox FDS — The Cardiox Shunt Detection system consists of a sensor placed in contact with the outer ear, similar to a finger probe used to detect oxygen levels in blood. Through an intravenous line, ICG (indocyanine green) at a dosage of 10 mg (2 mL of 5 mg/mL ICG solution) per test, is administered into the right or left antecubital fossa. The presence of ICG in the veins within the outer ear are detected, and the results are displayed on a monitor. All patients will also be evaluated with TCD and TEE for the presence of RTLS.

SUMMARY:
The CARDIOX Flow Detection System is designed to detect the presence of indocyanine green (ICG) dye in the blood and is being investigated to establish its efficacy in detecting the presence of right to left cardiac shunt (RTLS). The CARDIOX system will be compared against transesophageal echocardiography (TEE) for sensitivity and specificity, as well as transcranial doppler (TCD) for positive percent agreement and negative percent agreement.

ELIGIBILITY:
Inclusion Criteria:

* Eighteen (18) years of age or older
* Informed consent documentation understood and signed
* Planned or completed TEE study within the last 12 months

Exclusion Criteria:

* Subjects with a known allergy or sensitivity to Indocyanine Green Dye (ICG) or to Iodide Contrast Dye or Iodides
* Pregnant women or nursing mothers
* Subject unable or unwilling to understand and sign the informed consent
* Subject scheduled for radioactive iodine uptake test (Thyroid test) within 7 days of post screening
* Subjects that have poor renal function such as subjects on dialysis, subjects with a recent history of creatinine > 2.0 or subjects currently being followed by a nephrologist

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2011-04; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
To evaluate the Cardiox FDS system using TCD as a non-reference standard for positive percent agreement for accurately detecting a RTLS and negative percent agreement for accurately detecting the absence of RTLS | 1 day
To establish the safety of the Cardiox FDS device by tracking number of participants with adverse events related to Cardiox FDS | 1 day

SECONDARY OUTCOMES:
To evaluate the Cardiox FDS against TEE for sensitivity for the detection of RTLS and specificity for the detecting the absence of a shunt | 1 day

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - University of Alabama, Birmingham, Birmingham, Alabama
  - Heart and Vascular Center of Arizona, Phoenix, Arizona
  - UCLA Medical Center, Los Angeles, California
  - Tufts Medical Center, Boston, Massachusetts
  - Columbia University Medical Center, New York, New York
  - Riverside Methodist Hospital, Columbus, Ohio
  - Swedish Hospital, Seattle, Washington

REFERENCES:
- [Background] Karttunen V, Ventila M, Hillbom M, Salonen O, Haapaniemi H, Kaste M. Dye dilution and oximetry for detection of patent foramen ovale. Acta Neurol Scand. 1998 Apr;97(4):231-6. doi: 10.1111/j.1600-0404.1998.tb00643.x. PMID 9576637
- [Background] Spencer MP, Moehring MA, Jesurum J, Gray WA, Olsen JV, Reisman M. Power m-mode transcranial Doppler for diagnosis of patent foramen ovale and assessing transcatheter closure. J Neuroimaging. 2004 Oct;14(4):342-9. doi: 10.1177/1051228404268743. PMID 15358955